CLINICAL TRIAL: NCT03098888
Title: Bronchoalveolar Lavages in the Intensive Care Unit : Indications, Adverse Respiratory Effects, Contribution to Diagnosis and Therapy. A Multicenter, Prospective, Observational Study
Brief Title: Bronchoalveolar Lavages for Cytologic Assessment in Intensive Care Unit Patients
Acronym: REA-LBA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO cat III 2017-01; N° IDRCB 2017-A00306-47 (Other: French Government)
Record Dates: First submitted 2017-03-23; First posted 2017-04-04 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Lung Diseases; Intensive Care
Keywords: side effects; decision making; indications; risk factors
MeSH Terms: conditions — Lung Diseases | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bronchoalveolar lavage — bronchoalveolar lavages performed for cytological assessment in critically ill patients with lung diseases, intubated or not

SUMMARY:
Little is known about bronchoalveolar lavages performed for cytological assessment during bronchial fibroscopy in critically ill patients. Frequency of use, indications, actual contribution to diagnosis and therapeutic decision, and complications have not been extensively assessed.

The primary objective of this multi center, prospective, observational study is to describe the frequency of use of bronchoalveolar lavages for cytological assessement in critically ill patients, identify their indications, assess their contribution to diagnosis and therapeutic decisions, and estimate the frequency of induced respiratory events.

DETAILED DESCRIPTION:
Secondary objectives will be to

* assess the frequency of poor quality bronchoalveolar lavages (as defined by either more than 5% bronchial epithelial cell count to less than 50,000 alveolar cells per mL)
* assess the contribution of a given bronchoalveolar lavage to the diagnostic work up
* assess the contribution of a given bronchoalveolar lavage results to therapeutic decision
* assess the induced short term respiratory side effects
* identify risk factors for poor respiratory tolerance

ELIGIBILITY:
Inclusion Criteria:

* adult patient (> 18 yr-old) hospitalized in intensive care unit with acute and/or chronic lung disease that need bronchoalveolar lavage as part of routine diagnostic work up
* patient's or family consent

Exclusion Criteria:

* consent not obtained
* patient already included at previous bronchoalveolar lavage of during previous hospitalization
* absence of social security number
* age < 18yr
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients hospitalized in intensive care unit with acute and/or chronic lung disease that need bronchoalveolar lavage as part of the diagnostic work up
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
quality of performed bronchoalveolar lavage | 72 hours
  pathologists examining bronchoalveolar lavage specimen will classify bronchoalveolar lavage as "of poor quality" or of "good quality" based upon cytologic assessment: bronchial cell count (not more than 5%) and alveolar cell count (above 50,000/mL).
contribution to diagnosis and/or therapeutic decision | 72 hours
  Investigators will be ask to answer the following question: Did the bronchoalveolar lavage results contribute to diagnosis and/or therapeutic decision: Yes or No
frequency of use | 72 hours
  the frequency of use of bronchoalveolar lavage will be describe and expressed as the proportion of patients who underwent bronchoalveoalr lavage upon the total number of patients admitted in the recruiting intensive care units during the study period

SECONDARY OUTCOMES:
Evolution of respiratory rate | 24 hours
  respiratory rate will be assessed before the bronchoalveolar lavage and 8 times during the 24 hours following the bronchoalveolar lavage
Evolution of oxygen needs | 24 hours
  Oxygen needs, in L/min in patients under conventional nasal or facial oxygen therapy, or expressed in FiO2 in patients under nasal high flow oxygen or under invasive or noninvasive ventilation, will be recorded before bronchoalveolar lavage and 8 times during the following 24 hours.
Need of tracheal intubation | 24 hours
  Percentage of patients not intubated while undergoing bronchoalveolar lavage that will need intubation within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Toufik KAMEL, MD, Principal Investigator — CHR Orléans
Locations (16):
- France (16):
  - CHU d'ANGERS, Angers
  - CH d'ANGOULEME, Angoulême
  - CH Victor DUPOUY, Argenteuil
  - CHU de DIJON, Dijon
  - Hôpital RAYMOND POINCARE, Garches
  - CHD de VENDEE, La Roche-sur-Yon
  - CH de LA ROCHELLE, La Rochelle
  - Hopital de La Timone, Marseille
  - Hôpital Nord de Marseille, Marseille
  - CH de MONTAUBAN, Montauban
  - CHRU de NANTES, Nantes
  - CHR d'ORLEANS, Orléans
  - CHRU de POITIERS, Poitiers
  - CHU de STRASBOURG, Strasbourg
  - CHU de STRASBOURG NHC, Strasbourg
  - CHRU de TOURS, Tours

IPD SHARING:
Plan to Share IPD: No